CLINICAL TRIAL: NCT05248750
Title: Genetic, Microenvironmental, and Immunological Factors in Unresectable Pancreatic Ductal Adenocarcinoma
Status: Recruiting | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Guido Costamagna, Professor, Catholic University of the Sacred Heart
Other Study IDs: PDAC AIRC
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Pancreas Cancer
Keywords: pancreatic cancer; endoscopic ultrasound (EUS); personalized medicine
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) complexity, where genetic, stromal, and immunological factors all interact with each other, is responsible for the overall poor response of PDAC to chemotherapeutic agents, making this a lethal disease. The investigators hypothesize that: (i) dissection of genetic, stromal, and immunological factors on endoscopic ultrasound fine needle biopsy (EUS-FNB) tissue samples from unresectable PDAC patients' will allow to determine prognostic factors in this patient population; (ii) treatment response and acquisition of tumor chemotherapy resistance could be related to genetic heterogeneity between the primary and metastatic sites and alteration of the molecular profile under drug' selection pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to EUS with FNB for suspected pancreatic cancer unresectable or metastatic based on imaging findings
* Availability of biopsies obtained during EUS-FNB
* Histological diagnosis of pancreatic ductal adenocarcinoma of any stage
* Patients must be fit for chemotherapy administration
* They have to express their willingness to be followed up at our pancreatic high volume centers
* Age >18 and <80 years
* Able to sign informed consent

Exclusion Criteria:

* Histological diagnoses other than pancreatic ductal adenocarcinoma
* Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns consecutive individuals with a solid pancreatic lesion who will undergo diagnostic EUS-FNB over a 3 year period. Those with a histological diagnosis of PDAC will be enrolled in the study. Enrollment will include patients with unresectable disease, which can be divided in different stages, i.e. borderline resectable, locally advanced, and metastatic.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free-survival (PFS) | From date of enrollment assessed until death or up to 2 years
  To assess the impact of comprehensive genetic, stromal, and immunological factors on PFS defined as the time from the date of trial entry until disease progression or relapse.
Overall survival | From date of enrollment assessed until death or up to 2 years
  To assess the impact of comprehensive genetic, stromal, and immunological factors on Overall survival defined as the length of time (in days) between the treatment date and the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Larghi, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli
Locations (1):
- "Agostino Gemelli" Hospital, Catholic University of Sacred Heart, Rome, Lazio, Italy